## Title:

Simulation Training for Labor and Delivery Providers to Address HIV Stigma During Childbirth in Tanzania

NCT:

NCT05271903

**Document version:** 

November 6, 2020

## STATISTICAL DESIGN AND POWER

The goal of this study is to design and pilot test the MAMA intervention, a simulation training for labor and delivery providers that aims to reduce HIV stigma during the intrapartum period, improve the delivery of respectful maternity care for women living with HIV (WLHIV), and improve women's long-term HIV care engagement.

The primary outcome in the trial is respectful maternity care (RMC) scores of providers, comparing baseline and post-intervention. We will use summary statistics to describe participant characteristics and visualize trends over time. Mixed effect regressions will be used to assess the significance of observed changes from baseline to each follow-up timepoint, using means and 95% confidence intervals (CI).

As an R21 pilot study, it is not intended to be powered to be powered for a significant effect. Findings will help to calculate an effect size to properly power a future study.